CLINICAL TRIAL: NCT07061925
Title: A Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Multicenter, Dose-finding, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of ALC-2203 in Patients With Acute Bronchitis
Brief Title: To Evaluate the Efficacy and Safety of ALC-2203 in Patients With Acute Bronchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Arlico Pharm. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALC-2203-201
Record Dates: First submitted 2025-06-27; First posted 2025-07-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Bronchitis
Keywords: ALC-2203
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group 1 (Experimental)
  Interventions: Drug: ALC-2203-1
- Experimental Group 2 (Experimental)
  Interventions: Drug: ALC-2203-2
- Active Comparator Group (Active Comparator)
  Interventions: Drug: ALC-2203-AC
- Placebo Comparator Group (Placebo Comparator)
  Interventions: Drug: Placabo

INTERVENTIONS:
Drug: ALC-2203-1 — This group receives ALC-2203-1 and a placebo matching ALC-2203-AC, administered three times daily for 7 days.
  Arms: Experimental Group 1
Drug: ALC-2203-2 — This group receives ALC-2203-2 and a placebo matching ALC-2203-AC, administered three times daily for 7 days.
  Arms: Experimental Group 2
Drug: ALC-2203-AC — This group receives a placebo matching ALC-2203-1 or ALC-2203-2, and ALC-2203-AC, administered three times daily for 7 days.
  Arms: Active Comparator Group
Drug: Placabo — This group receives a placebo matching ALC-2203-1 or ALC-2203-2, and a placebo matching ALC-2203-AC, administered three times daily for 7 days.
  Arms: Placebo Comparator Group

SUMMARY:
A Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Multicenter, Dose-finding, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of ALC-2203 in Patients with Acute Bronchitis

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 19 years or older.
2. Patients diagnosed with acute bronchitis with:

   * A Bronchitis Severity Score (BSS) of ≥ 5 at Visit 2.
   * A sputum subscore of at least 1 at Visit 2.
3. Onset of acute bronchitis symptoms within 48 hours prior to Visit 2.
4. Patients who voluntarily agree to participate

Exclusion Criteria:

1. Patients who, in the opinion of the investigator, have severe respiratory diseases such as allergic asthma, chronic bronchitis, or asthma
2. Patients who are currently taking, or are expected to take during the study period, antitussive or expectorant medications containing agents such as codeine or dextromethorphan
3. Patients who have participated in another clinical trial within 4 weeks prior to screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Bronchitis Severity Score (BSS) at Day 7 | Baseline (Day 0) to Day 7
  The primary outcome measure is the change in total Bronchitis Severity Score (BSS) from baseline (Day 0) to Day 7 following administration of the investigational product.
  The BSS is a clinician-assessed tool used to evaluate five symptoms: cough, sputum, rales/rhonchi, chest pain during coughing, and dyspnea. Each symptom is scored on a scale from 0 to 4, yielding a total score ranging from 0 to 20.

SECONDARY OUTCOMES:
Change from baseline in Bronchitis Severity Score (BSS) at Day 4 | Baseline (Day 0) to Day 4
  The secondary outcome measure is the change in total Bronchitis Severity Score (BSS) from baseline (Day 0) to Day 4 following administration of the investigational product. The BSS is a clinician-assessed tool used to evaluate five symptoms: cough, sputum, rales/rhonchi, chest pain during coughing, and dyspnea. Each symptom is scored on a scale from 0 to 4, yielding a total score ranging from 0 to 20.
Change from baseline in individual BSS symptom scores at Day 4 and 7 | Baseline (Day 0) to Day 4 and Day 7
  Change in the individual symptom scores of BSS (cough, sputum, rales/rhonchi, chest pain during coughing, and dyspnea) from baseline (Day 0) to Day 4 and 7
Response rate based on BSS at Day 4 and Day 7 | Baseline (Day 0) to Day 4 and Day 7
  The proportion of participants who show a total BSS score <3 or a reduction of ≥7 points from baseline at Day 4 and Day 7
Investigator-assessed overall improvement and treatment effectiveness at Day 4 and 7 | Day 4 and Day 7
  Evaluation of the participant's overall improvement by the investigator using the Integrative Medicine Outcome Scale (IMOS). Treatment effectiveness is defined as an IMOS score of 4 ("major improvement") or 5 ("complete recovery")
Participant-reported overall satisfaction and satisfaction rate at Days 4 and 7 | Day 4 and Day 7
  Participant-reported overall satisfaction assessed using the Integrative Medicine Patient Satisfaction Scale (IMPSS). Satisfaction is defined as an IMPSS score of 4 ("satisfied") or 5 ("very satisfied")
Change from baseline in COAT total score at Day 4 and Day 7 | Baseline (Day 0) to Day 4 and Day 7
  Change in total score of the Cough Assessment Test (COAT), a participant-rated questionnaire assessing cough frequency, interference with daily life, sleep disturbance, fatigue, and hypersensitivity, each scored from 0 to 4 (total score: 0-20

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No